CLINICAL TRIAL: NCT06277167
Title: A Randomized, Double-Blind, Placebo-Controlled Phase-I Clinical Study to Evaluate the Tolerability, Safety and PK Profiles of Human Interferon Alfa 1b Inhalation Solution in Healthy Adult Subjects After Administration of Single Ascending Doses and Multiple Ascending Doses
Brief Title: A Phase I Study in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kexing Biopharm Co., Ltd. (Industry)
Collaborators: Guoxin Pharmaceutical Technology (Beijing) Co., Ltd. (Unknown); The Third Hospital of Changsha (Unknown); Beijing SSYP Data Technology Development Co.,Ltd. (Unknown); United-Power Pharma Tech（Shanghai）Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KXZY-GB05-101
Record Dates: First submitted 2024-02-02; First posted 2024-02-26 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Human interferon alfa 1b inhalation solution (SAD) (Experimental): Human interferon alfa 1b inhalation solution：200,000 IU, 600,000 IU, 1,200,000 IU, and 1,80,000 IU dose groups
  Interventions: Drug: Human interferon alfa 1b inhalation solution
- Human interferon alfa 1b inhalation solution placebo (SAD) (Placebo Comparator): Human interferon alfa 1b inhalation solution placebo ：200,000 IU, 600,000 IU, 1,200,000 IU, and 1,80,000 IU dose groups
  Interventions: Drug: Human interferon alfa 1b inhalation solution placebo
- Human interferon alfa 1b inhalation solution (MAD) (Experimental): Human interferon alfa 1b inhalation solution drug product：1,200,000 IU, and 1,80,000 IU dose groups
  Interventions: Drug: Human interferon alfa 1b inhalation solution
- Human interferon alfa 1b inhalation solution placebo (MAD) (Placebo Comparator): Human interferon alfa 1b inhalation solution placebo ：1,200,000 IU, and 1,80,000 IU dose groups
  Interventions: Drug: Human interferon alfa 1b inhalation solution placebo

INTERVENTIONS:
Drug: Human interferon alfa 1b inhalation solution — Participants will receive Human interferon alfa 1b inhalation solution orally for a single dose.
  Arms: Human interferon alfa 1b inhalation solution (SAD)
Drug: Human interferon alfa 1b inhalation solution placebo — Participants will receive Human interferon alfa 1b inhalation solution placebo orally for a single dose.
  Arms: Human interferon alfa 1b inhalation solution placebo (SAD)
Drug: Human interferon alfa 1b inhalation solution — Participants in the 1,200,000 IU and 1,800,000 IU dose groups will be given multiple consecutive doses after a single dose safety assessment, i.e. Human interferon alfa 1b inhalation solution administered by aerosol inhalation twice a day at the dose of the corresponding group, for 5 consecutive days respectively (only one morning dose on the last day, for a total of 10 doses during the study).
  Arms: Human interferon alfa 1b inhalation solution (MAD)
Drug: Human interferon alfa 1b inhalation solution placebo — Participants in the 1,200,000 IU and 1,800,000 IU dose groups will be given multiple consecutive doses after a single dose safety assessment, i.e. Human interferon alfa 1b inhalation solution placebo administered by aerosol inhalation twice a day at the dose of the corresponding group, for 5 consecutive days respectively (only one morning dose on the last day, for a total of 10 doses during the study).
  Arms: Human interferon alfa 1b inhalation solution placebo (MAD)

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled Phase-I Clinical Study to Evaluate the Tolerability, Safety and PK Profiles of Human interferon alfa 1b inhalation solution in Healthy Adult Subjects after Administration of Single Ascending Doses and Multiple Ascending Doses

DETAILED DESCRIPTION:
Primary objective:To evaluate the tolerability and safety of single and multiple aerosol inhalation of Human interferon alfa 1b inhalation solution in healthy adult subjects.

Secondary objectives: To evaluate the pharmacokinetic (PK) profiles of single and multiple aerosol inhalation of Human interferon alfa 1b inhalation solution in healthy adult subjects and to evaluate the immunogenicity of single and multiple aerosol inhalation of Human interferon alfa 1b inhalation solution in healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males or females aged 18-45 years;
2. Male body weight ≥45 kg, male body weight ≥50 kg, and body mass index (BMI): 19.0-26.0 kg/m2 (both inclusive), BMI =body weight (kg)/height 2 (m2);
3. The subjects voluntarily participate in the study and sign an informed consent form before the study.

Exclusion Criteria:

1. Subjects who participated in any clinical studies of drugs or took study drugs within 3 months prior to the administration of study drug;
2. Subjects who have undergone surgery within 3 months prior to screening or who plan to undergo surgery during the study or who have undergone surgery that would affect the absorption, distribution, metabolism, and excretion of drugs; subjects with a previous history of diseases of cardiovascular system, blood and lymphatic system, respiratory system, urinary system, endocrine, immune, mental and nervous system (such as epilepsy) that are clinically significant;
3. Subjects with a history of respiratory system diseases, such as acute exacerbation of chronic obstructive pulmonary disease, pulmonary fibrosis, pulmonary hypertension, pulmonary edema, pulmonary interstitial disease, bronchial asthma, paradoxical bronchospasm, or throat ulcer and edema, or subjects with previous surgery of throat, trachea/bronchi and lung, or subjects with upper and lower respiratory tract infection and acute sinusitis caused by virus or bacteria within the 4 weeks prior to the use of study drug that are clinically significant or render them unsuitable to participate in the study in the opinion of the investigator;
4. Subjects with ocular diseases or thyroid-related diseases that are clinically significant or render them unsuitable to participate in the study in the opinion of the investigator;
5. Subjects with a history of drug allergy (antibiotics, interferon products, etc.), or a specific history of allergy (asthma, urticaria, eczema, etc.), or allergic constitution (such as allergy to two or more drugs, food, pollen, etc.);
6. Subjects who cannot tolerate aerosol inhalation;
7. Subjects who have used any prescription drugs, over-the-counter drugs, Chinese herbal medicines, or vitamins within14 days prior to screening;
8. Subjects who have received vaccine within 4 weeks prior to the first dose, or subjects who plan to receive vaccine within 4 weeks after the last dose;
9. Subjects who have had non-physiological blood loss of ≥300 mL within 3 months before the first dose (including trauma, blood collection, blood donation); or subjects who plan to donate blood during the study or within 30 days after the last dose;
10. Subjects who have had a history of drug use or abuse within 6 months prior to screening;
11. Subjects who have smoked within 3 months prior to screening, or who cannot stop using any tobacco products during the study;
12. Subjects who have consumed more than 14 glasses of alcohol per week (1 glass =150 mL wine, or 360 mL beer, or 45 mL spirits) within 3 months prior to screening;
13. Subjects who cannot tolerate venipuncture for blood collection or have potential blood collection difficulties, or subjects who feel dizzy and sick at the sight of blood or needle;
14. Subjects who have special requirements for diet and cannot follow a standardized diet;
15. Subjects who have a birth plan, or are unable to voluntarily take effective contraceptive measures, or have a sperm/egg donation plan during the study period and within 3 months after the last dose; female subjects who are pregnant or lactating;
16. Subjects with clinically significant abnormalities on physical examinations, electrocardiograms, vital signs, chest X-rays, lung function, and laboratory tests (as judged by the clinician);
17. Pulmonary function test: subjects with measured/predicted FEV1 ≤80% or FVC≤ 80% of expected value;
18. Subjects who have positive urine nicotine test results;
19. Subjects who have positive urine drug test results;
20. Subjects who have positive alcohol breath results;
21. Subjects who cannot use aerosol device correctly or who do not pass the aerosol dosing training;
22. Subjects who cannot complete this study due to other reasons, or subjects who are unsuitable to participate in this clinical study due to other various reasons;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2023-01-07 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
TEAEs | Day 1 up to 29 or Day 1 up to 32
  The adverse events and incidence of treatment-emergent adverse events(TEAEs)
(ADRs) | Day 1 up to 29 or Day 1 up to 32
  The adverse events and incidence of adverse drug reactions (ADRs)
(SAE) | Day 1 up to 29 or Day 1 up to 32
  The adverse events and incidence of serious adverse events (SAE)
TEAEs that lead to subject discontinuation from the study | Day 1 up to 29 or Day 1 up to 32
  The adverse events and incidence of TEAEs that lead to subject discontinuation from the study

SECONDARY OUTCOMES:
Cmax After a Single Dose of GB05 Drug Product | Day 1 up to 3
  The maximum concentration (Cmax) of GB05 Drug Product
Tmax After a Single Dose of GB05 Drug Product | Day 1 up to 3
  The maximum concentration (Tmax) of GB05 Drug Product
AUC0-t and AUC0-inf After a Single Dose of GB05 Drug Product | Day 1 up to 3
  The area under the concentration-time curve (AUC0-t and AUC0-inf) of GB05 Drug Product.
t1/2 After a Single Dose of GB05 Drug Product | Day 1 up to 3
  The elimination half-life (t1/2) of GB05 Drug Product
Ke After a Single Dose of GB05 Drug Product | Day 1 up to 3
  The elimination rate constant (Ke) of GB05 Drug Product
Vd After a Single Dose of GB05 Drug Product | Day 1 up to 3
  The apparent distribution volume (Vd) of GB05 Drug Product.
MRT After a Single Dose of GB05 Drug Product | Day 1 up to 3
  The average residence time (MRT) of GB05 Drug Product
CL After a Single Dose of GB05 Drug Product | Day 1 up to 3
  The clearance rate (CL) of GB05 Drug Product
Cmax,ss After Multiple Doses of GB05 Drug Product | Day 1 up to 10
  The maximum concentration at steady state (Cmax,ss) of GB05 Drug Product
Cmin,ss After Multiple Doses of GB05 Drug Product | Day 1 up to 10
  The minimum concentration at steady state (Cmin,ss) of GB05 Drug Product
Css_av After Multiple Doses of GB05 Drug Product | Day 1 up to 10
  The average steady-state plasma concentration (Css_av) of GB05 Drug Product
DF After Multiple Doses of GB05 Drug Product | Day 1 up to 10
  The degree of fluctuation in the concentration during the dosing interval (DF) of GB05 Drug Product
(Cmax,ss-Cmin,ss)/Cmin,ss After Multiple Doses of GB05 Drug Product | Day 1 up to 10
  The fluctuation amplitude [(Cmax,ss-Cmin,ss)/Cmin,ss] of GB05 Drug Product
ADA | Day 1 up to 29 or Day 1 up to 32
  The Number and Percentage of Participants of anti-drug antibody (ADA)
NAb | Day 1 up to 29 or Day 1 up to 32
  The Number and Percentage of Participants of neutralizing antibody (NAb).

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Hospital of Changsha, Changsha, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peng H, Zhang W, Lin Y, Li H, Qin S. Safety, Tolerability, and Pharmacokinetics of Nebulized GB05-Human IFNalpha1b Inhalation Solution: A Randomized, Placebo-Controlled, Dose-Escalation Phase I Study in Healthy Chinese Adult Volunteers. Infect Dis Ther. 2024 Sep;13(9):2053-2070. doi: 10.1007/s40121-024-01024-y. Epub 2024 Aug 4. PMID 39097549